CLINICAL TRIAL: NCT00043381
Title: A Randomized, Open-label, Phase III Trial of Decitabine (5-aza-2'Deoxycytidine) Versus Supportive Care in Adults With Advanced-stage Myelodysplastic Syndrome
Brief Title: Decitabine Versus Supportive Care in Adults With Advanced-stage MDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: David S. Smith, Vice President-Regulatory and Quality Assurance, SuperGen, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-0007; NCT00022061 (obsolete NCT alias)
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; MDS; chronic myelomonocytic leukemia; CMML; decitabine; 5-aza-2'deoxycytidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine (5-aza-2'deoxycytidine)

SUMMARY:
To compare the safety and efficacy profiles of decitabine to those of supportive care in adults with advanced-stage myelodysplastic syndrome (MDS)

DETAILED DESCRIPTION:
This experimental (investigational) study is intended to answer the question of whether decitabine is any better than supportive care alone in delaying progression (worsening) of the disease, prolonging survival or improving the overall quality of life for MDS patients who are not candidates for bone marrow transplant (BMT).

ELIGIBILITY:
Inclusion:

* MDS (de novo or secondary) fitting any of the recognized French-American-British, FAB, classifications or chronic myelomonocytic leukemia (CMML) with WBC < 12,000/mm3, AND International Prognostic Scoring System (IPSS) >/= 0.5 as determined by CBC, bone marrow assessment and bone marrow cytogenetics within 30 days of randomization
* 18 years or older
* Female patients of child-bearing potential must have a negative serum hCG within 24 hours prior to randomization, must practice a medically approved method of birth control for the past 30 days, and agree to continue this practice for the trial duration and must not be breast-feeding
* ECOG or WHO performance status of 0-2
* Written informed consent
* Normal renal and hepatic function (creatinine </= 2 mg/dL, bilirubin </= 1.5 mg/dL, SGPT </= 2 times the upper limit of normal range)

Exclusion:

* Acute Myeloid Leukemia (AML) (>/=30% bone marrow blasts) or other progressive malignant disease
* Patients must have recovered from the toxic effects of prior therapy and must be off all chemotherapy for a minimum of 4 weeks prior to study entry to the protocol (a minimum of six weeks for prior nitrosoureas and bone marrow transplantation)
* Ongoing treatment with androgenic hormones, danazol, colony-stimulating factors, or other agents used to treat MDS within 7 days of study initiation.
* Administration of any investigational agent within the 30 days preceding study initiation.
* Uncontrolled cardiac disease or congestive heart failure
* Uncontrolled restrictive or obstructive pulmonary disease
* Active viral or bacterial infection
* Superimposed autoimmune hemolytic anemia or thrombocytopenia
* Known positive serology for HIV
* Mental illness or other condition preventing full cooperation with the treatment and monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-04; Primary Completion 2002-11 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - City of Hope National Medical Center, Duarte, California
  - Scripps Clinic, Escondido, California
  - Loma Linda Univ. Cancer Center, Loma Linda, California
  - Univ. California San Francisco Medical School, San Francisco, California
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - James A. Haley Veteran's Hospital, Tampa, Florida
  - Rush Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - New England Medical Center Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - VA Medical Center, Minneapolis, Minnesota
  - Washington Univ. School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Memphis Cancer Center, Memphis, Tennessee
  - SW Regional Cancer Center (dba Central Texas Oncology Associates), Austin, Texas
  - Texas Oncology, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Jabbour E, Kantarjian H, O'Brien S, Kadia T, Malik A, Welch MA, Teng A, Cortes J, Ravandi F, Garcia-Manero G. Retrospective analysis of prognostic factors associated with response and overall survival by baseline marrow blast percentage in patients with myelodysplastic syndromes treated with decitabine. Clin Lymphoma Myeloma Leuk. 2013 Oct;13(5):592-6. doi: 10.1016/j.clml.2013.05.004. Epub 2013 Jun 20. PMID 23790798
- [Derived] Jabbour E, Garcia-Manero G, Ravandi F, Faderl S, O'Brien S, Fullmer A, Cortes JE, Wierda W, Kantarjian H. Prognostic factors associated with disease progression and overall survival in patients with myelodysplastic syndromes treated with decitabine. Clin Lymphoma Myeloma Leuk. 2013 Apr;13(2):131-8. doi: 10.1016/j.clml.2012.11.001. Epub 2012 Dec 21. PMID 23260600